CLINICAL TRIAL: NCT04350359
Title: Transcutaneous Tibial Nerve Stimulation for Spinal Cord Injury Neurogenic Bladder
Acronym: TTNS1yr
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: MedStar National Rehabilitation Network (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Argyrios Stampas, MD, Spinal Cord Injury Medicine Research Director, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-19-0756
Record Dates: First submitted 2020-04-02; First posted 2020-04-17 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries
Keywords: electric stimulation; SCI; spinal cord injury; neurogenic bladder
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: A prospective, double-blinded, randomized trial.
Who Masked: Investigator
Masking Description: Subjects will be randomized to either Variable or fixed-dose (2:1) using a block size of 6 and stratified based on complete/incomplete SCI to ensure the equal allocation of the most severely injured in the two groups. The PI and investigators will be blinded to randomization and treatment allocation, managed by the research assistant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Variable-dose TTNS Protocol 5 x week (Active Comparator): TTNS protocol: Electrodes 2 inch by 2 inch will be placed according to anatomic landmarks, with the negative electrode behind the internal malleolus and the positive electrode 10cm superior to the negative electrode, verified with rhythmic flexion of the toes secondary to stimulation of the flexor digitorum and hallicus brevis. The intensity level will be set to the amperage immediately under the threshold for motor contraction. If there is no contraction seen, patients will be excluded. In addition, if the patient perceives pain, the intensity will be lowered until comfortable. Stimulation frequency of 20 Hz and pulse width of 200ms in continuous mode will be used.
  All participants will be instructed to use the device for 30 minutes, 5 days per week for the first 4 months post-sci.
  Interventions: Device: Variable-dose TTNS Protocol 5 x week
- Fixed-dose TTNS protocol (Active Comparator): Fixed-dose protocol: Toe flexion will be attempted, as in the TTNS protocol. Then the stimulation will be reduced to 1 mA for 30 minutes.
  Both variable-dose TTNS and fixed-dose TTNS protocol participants will be instructed to use the device for 30 minutes, 5 days per week.
  Interventions: Device: Fixed-dose TTNS Protocol
- Variable-dose TTNS Protocol 2 x week (Active Comparator): At the 4 month CMG, subjects initially randomized into the variable dose protocol of 2 x weekly will start doing so for the remainder of the study.
  Interventions: Device: Variable-dose TTNS Protocol 2 x week

INTERVENTIONS:
Device: Variable-dose TTNS Protocol 5 x week — Electrodes 2 inch by 2 inch will be placed according to anatomic landmarks, with the negative electrode behind the internal malleolus and the positive electrode 10cm superior to the negative electrode, verified with rhythmic flexion of the toes secondary to stimulation of the flexor digitorum and hallicus brevis. The intensity level will be set to the amperage immediately under the threshold for motor contraction. If there is no contraction seen, patients will be excluded. In addition, if the patient perceives pain, the intensity will be lowered until comfortable. Stimulation frequency of 20 Hz and pulse width of 200ms in continuous mode will be used.
  Arms: Variable-dose TTNS Protocol 5 x week
Device: Fixed-dose TTNS Protocol — Toe flexion will be attempted, as in the TTNS protocol. Then the stimulation will be reduced to 1 mA for 30 minutes. This will continue at 5x weekly until 1-year post-injury.
  Arms: Fixed-dose TTNS protocol
Device: Variable-dose TTNS Protocol 2 x week — At the 4 month CMG, subjects initially randomized into the variable dose protocol of 2 x weekly will start doing so for the remainder of the study.
  Arms: Variable-dose TTNS Protocol 2 x week

SUMMARY:
The purpose of this study is to determine if electric stimulation to the leg, called transcutaneous tibial nerve stimulation (TTNS), can improve bladder outcomes in acute spinal cord injury.

DETAILED DESCRIPTION:
The purpose of this study is to see how well TTNS works at preventing incontinence in people with paraplegia from SCI that perform intermittent catheterization to empty their bladder. This study will compare the effectiveness of TTNS at 2 doses, fixed-dose and variable-dose. It will also evaluate the frequency of use, 2 days weekly compared to 5 days weekly.

Based on our pilot trials, tibial nerve stimulation protocols use submotor current intensity with a duration of 200 µs and a frequency of 20Hz. The experimental group will use a submotor "variable dose." The fixed-dose group will use submotor at current intensity at 1mA and designated as "fixed-dose."

TTNS will be used 5 days weekly, per our pilot trial. At 4-months post-SCI, the subject will be instructed to switch to 2x daily if he or she was randomized into the variable dose group of 2 days weekly and thus continue to doing so for the remainder of study participation. Because there is support in the literature for reduced doses of tibial nerve stimulation required for maintenance (1-3x weekly), the RCT includes this frequency comparison arm. All subjects will continue for 1-year post-SCI.

Additionally, we are collecting surveys to help identify characteristics of people (resilience and confidence) and adherence to medication and TTNS use throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Traumatic or non-traumatic SCI
* Admitted to inpatient rehabilitation within 6 weeks
* T9 level of injury and above who are at greatest risk of morbid NGB
* Regionally located to allow follow-up
* English or Spanish speaking

Exclusion Criteria:

* History of genitourinary diagnoses (i.e. prostate hypertrophy, overactive bladder, cancer, etc.)
* History of central nervous system disorder (i.e. prior SCI, stroke, brain injury, Parkinson's disease, MS, etc.)
* History of peripheral neuropathy
* pre-SCI symptoms of peripheral neuropathy (numbness and/or tingling in feet, sharp/jabbing/burning pain in feet, sensitivity to touch, lack of coordination, muscle weakness, etc.)
* Pregnancy
* Known injury to the lumbosacral spinal cord or plexus, or pelvis with associated neuropathy
* concern for tibial nerve pathway injury
* absence of toe flexion or autonomic dysreflexia during electric stimulation test
* Potential for progressive SCI including neurodegenerative SCI, ALS, cancer myelopathy, Multiple sclerosis, transverse myelitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Maintained bladder capacity as assessed by the Urodynamics study measured in ml | Baseline
  we expect bladder capacity to be maintained in those with effective TTNS
Maintained bladder capacity as assessed by the Urodynamics study measured in ml | 4 months post SCI
  we expect bladder capacity to be maintained in those with effective TTNS
Prolonged sensation with bladder filling as assessed by the Urodynamics study measured in ml | Baseline
  Evidence of TTNS mechanism expected in those with effective TTNS
Prolonged sensation with bladder filling as assessed by the Urodynamics study measured in ml | 4 months post SCI
  Evidence of TTNS mechanism expected in those with effective TTNS
Prolonged sensation with bladder filling as assessed by the Urodynamics study measured in ml | 1 year post SCI
  Evidence of TTNS mechanism expected in those with effective TTNS
Change in bladder pathology from baseline presence of detrusor overactivity and DSD as assessed by the urodynamics study at 4 months. | Baseline, 4 months
  Reduced bladder pathology (presence of detrusor overactivity and DSD) in those with effective bladder neuromodulation based on change in urodynamic studies at baseline and 4-months
Change in bladder pathology from 4 month presence of detrusor overactivity and DSD as assessed by the urodynamics study at 1 year post SCI. | 4 months and 1 year post SCI
  Reduced bladder pathology (presence of detrusor overactivity and DSD) in those with effective bladder neuromodulation based on the change in urodynamic studies at 4 months and 1-year

SECONDARY OUTCOMES:
Evidence of improved quality of life in those with effective bladder neuromodulation based on Incontinence Quality of Life (I-QOL) survey | At discharge which could be up to 4 week from admission, 4-months post injury and at 1 year post injury.
  Comparing I-QOL upon discharge from rehabilitation, 4-months post-injury and 1-year post-injury using incontinence QOL (I-QOL) survey, between and within both arms of the study
Evidence of improved quality of life in those with effective bladder neuromodulation based on Neurogenic Bladder Symptom Score (NBSS) | Prior to discharge which could be up to 4 weeks from admission, monthly until 1 year post injury.
  Changes in Neurogenic Bladder Symptom Scores. The total score can range from 0 (no symptoms at all) to 74 (maximum symptoms) where a lower score indicates a better outcome.
Evidence of improved quality of life in those with effective bladder neuromodulation based on frequency of catheterization and voiding volumes | 2 days at the end of each month for 1 year.
  Maintaining frequency of catheterization (count per day) and volumes per void (ml per collection)

CONTACTS AND LOCATIONS:
Overall Officials: Argyrios Stampas, MD, Principal Investigator — UTHealth and TIRR Mermorial Hermann; Suzanne Groah, MD, Principal Investigator — MedStar National Rehabilitation Hospital
Locations (2):
- United States (2):
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia
  - TIRR Memorial Hermann Research Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackery A, Tator C, Krassioukov A. A global perspective on spinal cord injury epidemiology. J Neurotrauma. 2004 Oct;21(10):1355-70. doi: 10.1089/neu.2004.21.1355. PMID 15672627
- [Background] Weld KJ, Dmochowski RR. Association of level of injury and bladder behavior in patients with post-traumatic spinal cord injury. Urology. 2000 Apr;55(4):490-4. doi: 10.1016/s0090-4295(99)00553-1. PMID 10736489
- [Background] Stohrer M, Blok B, Castro-Diaz D, Chartier-Kastler E, Del Popolo G, Kramer G, Pannek J, Radziszewski P, Wyndaele JJ. EAU guidelines on neurogenic lower urinary tract dysfunction. Eur Urol. 2009 Jul;56(1):81-8. doi: 10.1016/j.eururo.2009.04.028. Epub 2009 Apr 21. PMID 19403235
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Chaabane W, Guillotreau J, Castel-Lacanal E, Abu-Anz S, De Boissezon X, Malavaud B, Marque P, Sarramon JP, Rischmann P, Game X. Sacral neuromodulation for treating neurogenic bladder dysfunction: clinical and urodynamic study. Neurourol Urodyn. 2011 Apr;30(4):547-50. doi: 10.1002/nau.21009. PMID 21488095
- [Background] Chen G, Liao L, Li Y. The possible role of percutaneous tibial nerve stimulation using adhesive skin surface electrodes in patients with neurogenic detrusor overactivity secondary to spinal cord injury. Int Urol Nephrol. 2015 Mar;47(3):451-5. doi: 10.1007/s11255-015-0911-6. Epub 2015 Jan 22. PMID 25609546
- [Background] del Popolo G, Mencarini M, Nelli F, Lazzeri M. Controversy over the pharmacological treatments of storage symptoms in spinal cord injury patients: a literature overview. Spinal Cord. 2012 Jan;50(1):8-13. doi: 10.1038/sc.2011.110. Epub 2011 Nov 1. PMID 22042300
- [Background] Canbaz Kabay S, Kabay S, Mestan E, Cetiner M, Ayas S, Sevim M, Ozden H, Karaman HO. Long term sustained therapeutic effects of percutaneous posterior tibial nerve stimulation treatment of neurogenic overactive bladder in multiple sclerosis patients: 12-months results. Neurourol Urodyn. 2017 Jan;36(1):104-110. doi: 10.1002/nau.22868. Epub 2015 Sep 9. PMID 26352904
- [Background] Sirls ER, Killinger KA, Boura JA, Peters KM. Percutaneous Tibial Nerve Stimulation in the Office Setting: Real-world Experience of Over 100 Patients. Urology. 2018 Mar;113:34-39. doi: 10.1016/j.urology.2017.11.026. Epub 2017 Nov 28. PMID 29196071
- [Background] Fougere RJ, Currie KD, Nigro MK, Stothers L, Rapoport D, Krassioukov AV. Reduction in Bladder-Related Autonomic Dysreflexia after OnabotulinumtoxinA Treatment in Spinal Cord Injury. J Neurotrauma. 2016 Sep 15;33(18):1651-7. doi: 10.1089/neu.2015.4278. Epub 2016 Apr 13. PMID 26980078
- [Background] Sievert KD, Amend B, Gakis G, Toomey P, Badke A, Kaps HP, Stenzl A. Early sacral neuromodulation prevents urinary incontinence after complete spinal cord injury. Ann Neurol. 2010 Jan;67(1):74-84. doi: 10.1002/ana.21814. PMID 20186953
- [Background] de Seze M, Raibaut P, Gallien P, Even-Schneider A, Denys P, Bonniaud V, Game X, Amarenco G. Transcutaneous posterior tibial nerve stimulation for treatment of the overactive bladder syndrome in multiple sclerosis: results of a multicenter prospective study. Neurourol Urodyn. 2011 Mar;30(3):306-11. doi: 10.1002/nau.20958. Epub 2011 Feb 8. PMID 21305588
- [Background] McDonald JW 3rd, Sadowsky CL, Stampas A. The changing field of rehabilitation: optimizing spontaneous regeneration and functional recovery. Handb Clin Neurol. 2012;109:317-36. doi: 10.1016/B978-0-444-52137-8.00020-6. PMID 23098722
- [Background] Stampas A, Tansey KE. Spinal cord injury medicine and rehabilitation. Semin Neurol. 2014 Nov;34(5):524-33. doi: 10.1055/s-0034-1396006. Epub 2014 Dec 17. PMID 25520024
- [Background] Stampas A, York HS, O'Dell MW. Is the Routine Use of a Functional Electrical Stimulation Cycle for Lower Limb Movement Standard of Care for Acute Spinal Cord Injury Rehabilitation? PM R. 2017 May;9(5):521-528. doi: 10.1016/j.pmrj.2017.03.005. No abstract available. PMID 28526124
- [Background] Stampas A, Korupolu R, Zhu L, Smith CP, Gustafson K. Safety, Feasibility, and Efficacy of Transcutaneous Tibial Nerve Stimulation in Acute Spinal Cord Injury Neurogenic Bladder: A Randomized Control Pilot Trial. Neuromodulation. 2019 Aug;22(6):716-722. doi: 10.1111/ner.12855. Epub 2018 Oct 3. PMID 30284350
- [Background] Sanford MT, Suskind AM. Neuromodulation in neurogenic bladder. Transl Androl Urol. 2016 Feb;5(1):117-26. doi: 10.3978/j.issn.2223-4683.2015.12.01. PMID 26904417
- [Background] Stampas A, Gustafson K, Korupolu R, Smith C, Zhu L, Li S. Bladder Neuromodulation in Acute Spinal Cord Injury via Transcutaneous Tibial Nerve Stimulation: Cystometrogram and Autonomic Nervous System Evidence From a Randomized Control Pilot Trial. Front Neurosci. 2019 Feb 19;13:119. doi: 10.3389/fnins.2019.00119. eCollection 2019. PMID 30837835
- [Background] Finazzi Agro E, Campagna A, Sciobica F, Petta F, Germani S, Zuccala A, Miano R. Posterior tibial nerve stimulation: is the once-a-week protocol the best option? Minerva Urol Nefrol. 2005 Jun;57(2):119-23. English, Italian. PMID 15951736
- [Background] Manriquez V, Guzman R, Naser M, Aguilera A, Narvaez S, Castro A, Swift S, Digesu GA. Transcutaneous posterior tibial nerve stimulation versus extended release oxybutynin in overactive bladder patients. A prospective randomized trial. Eur J Obstet Gynecol Reprod Biol. 2016 Jan;196:6-10. doi: 10.1016/j.ejogrb.2015.09.020. Epub 2015 Oct 20. PMID 26645117
- [Background] Gaziev G, Topazio L, Iacovelli V, Asimakopoulos A, Di Santo A, De Nunzio C, Finazzi-Agro E. Percutaneous Tibial Nerve Stimulation (PTNS) efficacy in the treatment of lower urinary tract dysfunctions: a systematic review. BMC Urol. 2013 Nov 25;13:61. doi: 10.1186/1471-2490-13-61. PMID 24274173
- [Background] Dubeau CE. The aging lower urinary tract. J Urol. 2006 Mar;175(3 Pt 2):S11-5. doi: 10.1016/S0022-5347(05)00311-3. PMID 16458733
- [Background] Welk B, Lenherr S, Elliott S, Stoffel J, Presson AP, Zhang C, Myers JB. The Neurogenic Bladder Symptom Score (NBSS): a secondary assessment of its validity, reliability among people with a spinal cord injury. Spinal Cord. 2018 Mar;56(3):259-264. doi: 10.1038/s41393-017-0028-0. Epub 2017 Nov 29. PMID 29184133
- [Background] Schurch B, Denys P, Kozma CM, Reese PR, Slaton T, Barron R. Reliability and validity of the Incontinence Quality of Life questionnaire in patients with neurogenic urinary incontinence. Arch Phys Med Rehabil. 2007 May;88(5):646-52. doi: 10.1016/j.apmr.2007.02.009. PMID 17466735
- [Background] Bothig R, Fiebag K, Thietje R, Faschingbauer M, Hirschfeld S. Morbidity of urinary tract infection after urodynamic examination of hospitalized SCI patients: the impact of bladder management. Spinal Cord. 2013 Jan;51(1):70-3. doi: 10.1038/sc.2012.107. Epub 2012 Sep 11. PMID 22964752
- [Background] Pannek J, Nehiba M. Morbidity of urodynamic testing in patients with spinal cord injury: is antibiotic prophylaxis necessary? Spinal Cord. 2007 Dec;45(12):771-4. doi: 10.1038/sj.sc.3102114. Epub 2007 Aug 21. PMID 17710104
- [Background] Street JT, Noonan VK, Cheung A, Fisher CG, Dvorak MF. Incidence of acute care adverse events and long-term health-related quality of life in patients with TSCI. Spine J. 2015 May 1;15(5):923-32. doi: 10.1016/j.spinee.2013.06.051. Epub 2013 Aug 24. PMID 23981816
- [Background] Montgomerie JZ. Infections in patients with spinal cord injuries. Clin Infect Dis. 1997 Dec;25(6):1285-90; quiz 1291-2. doi: 10.1086/516144. No abstract available. PMID 9431366